CLINICAL TRIAL: NCT07038785
Title: A Double Blind Observational Study to Validate the SpotitEarly Test for the Detection of Breast Cancer (The PINK Study)
Brief Title: Identification of Breast Cancer in Breath Samples Using Trained Detection Dogs
Acronym: PINK
Status: Recruiting | Type: Observational
Sponsor: SpotitEarly (Industry)
Collaborators: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Other Study IDs: P-0001; Pro2024-0383 (Other: Hackensack Meridian Health)
Record Dates: First submitted 2025-06-11; First posted 2025-06-26 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Screening; Breath Samples; Cancer Detection
MeSH Terms: conditions — Breast Neoplasms | interventions — Breath Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Exhaled breath samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Target Population Arm: Women scheduled for routine breast cancer screening by mammography/ultrasound/magnetic resonance imaging
  Interventions: Diagnostic Test: Breath test
- Enriched Arm: Women scheduled for breast biopsy with a Breast Imaging and Reporting Data System (BI-RADS®) score of 4B or above
  Interventions: Diagnostic Test: Breath test

INTERVENTIONS:
Diagnostic Test: Breath test — Breath sample collection using a sample collection kit

SUMMARY:
The goal of this study is to find out whether a system that uses trained detection dogs and artificial intelligence (AI) can identify breast cancer from a person's breath. Women who are scheduled to have routine breast cancer screening, such as a mammogram, ultrasound, or a biopsy for a possible cancer, will be invited to take part. Participants will be asked to breathe into a surgical mask to collect a breath sample.

The mask will be sent to a special laboratory, where trained dogs and an AI-based system will check the sample for signs of breast cancer. The results from the dogs and AI will be compared to the actual results from the medical screening or biopsy to see how accurate the system is at detecting breast cancer.

ELIGIBILITY:
INCLUSION CRITERIA FOR ARM 1 (TARGET POPULATION ARM)

1. Capable of giving informed consent for self, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
2. Assigned female at birth.
3. 40 years of age and above OR
4. Between 18 and 39 years of age (inclusive) and a carrier of germline pathogenic variants associated with high risk for breast cancer: BRCA1, BRCA2, PTEN, TP53, CDH1, or STK11 ATM, CHEK2, BARD1, RAD51D, RAD51C, PALB2, OR
5. Between 18 and 39 years of age (inclusive) with a family history of breast or ovarian cancer involving at least one first or two second-degree relatives who were diagnosed with breast or ovarian cancer before the age of 50 years.
6. Scheduled for routine annual breast cancer screening (Mammogram, Ultrasound and MRI)

INCLUSION CRITERIA FOR ARM 2 (ENRICHED ARM)

1. Capable of giving informed consent for self, which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.
2. Assigned female at birth.
3. 40 years of age and above. OR
4. Between 18 and 39 years of age (inclusive) and a carrier of germline pathogenic variants associated with high risk for breast cancer: BRCA1, BRCA2, PTEN, TP53, CDH1, or STK11 ATM, CHEK2, BARD1, RAD51D, RAD51C, PTEN , PALB2 OR
5. Between 18 and 30 years of age (inclusive) with a family history of breast or ovarian cancer involving at least one first or two second-degree relatives who were diagnosed with breast or ovarian cancer before the age of 35 years.
6. BI-RADS® score of 4B.
7. Scheduled for breast biopsy.

EXCLUSION CRITERIA (BOTH STUDY ARMS)

1. Had cancer within the past year. Individuals who underwent surgical removal of cancerous non-metastatic skin lesions can be recruited.
2. Has received any cancer treatments within the past year.
3. Has participated in another clinical study in the past 30 days.
4. Had bilateral mastectomy for breast cancer or for preventive reasons related to breast cancer.
5. Had a medical procedure in the chest cavity and/or airways within the past 2 weeks which may interfere with the ability to provide a normal breath sample as required by the protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All eligible subjects who are seen at the medical center/study site for their breast cancer screening and biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 1204 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Test Performance Evaluation | 24 months
  The test performance will be determined by analysis of the sensitivity and the specificity of the primary endpoint sample set, where sensitivity is the number of participants with a true positive result divided by the number of participants with a positive clinical diagnosis (positive biopsy), and specificity is the number of participants with a true negative result divided by the number of participants with a negative clinical diagnosis.

SECONDARY OUTCOMES:
Test Performance Evaluation in different subgroups | 24 months
  Sensitivity and specificity of the SpotitEarly test will be measured and compared in each of the subgroups:
  * Age: under 40, 40-49, 50-64, 65 and older.
  * Race: White, Black/African American, Asian.
  * Ethnicity: hispanic vs. non hispanic
  * Germline pathogenic variant carriers associated with high risk for breast cancer versus non carriers.
  * Smoking status: smokers versus nonsmokers.
  * Women with type-2 diabetes versus not diagnosed with type-2 diabetes Sensitivity is the number of participants with a true positive result divided by the number of participants with a positive clinical diagnosis (positive biopsy). Specificity is the number of participants with a true negative result divided by the number of participants with a negative clinical diagnosis.
Test Performance in early-stage cancer | 24 months
  To evaluate the performance (sensitivity and specificity) of the SpotitEarly test in detecting early-stage breast cancer (stages 0-2).
  Sensitivity is the number of participants with a true positive result divided by the number of participants with a positive clinical diagnosis (positive biopsy). Specificity is the number of participants with a true negative result divided by the number of participants with a negative clinical diagnosis.
Test Performance in the clinic vs. at patients' home | 24 months
  To evaluate the performance (sensitivity and specificity, as described in 3.4) of the SpotitEarly test over samples provided by participants at their home.
  Sensitivity is the number of participants with a true positive result divided by the number of participants with a positive clinical diagnosis (positive biopsy). Specificity is the number of participants with a true negative result divided by the number of participants with a negative clinical diagnosis.
Effect of psychological impacts on performance in the enriched arm | 12 months
  To assess whether the performance (sensitivity and specificity) of the SpotitEarly test is affected by the subject's psychological impacts (anxiety is assumed for all arm 2 subjects who are undergoing a biopsy).
  Sensitivity is the number of participants with a true positive result divided by the number of participants with a positive clinical diagnosis (positive biopsy). Specificity is the number of participants with a true negative result divided by the number of participants with a negative clinical diagnosis.

CONTACTS AND LOCATIONS:
Locations (5):
- Hackensack Meridian Health, Totowa, New Jersey, United States
- Israel (4):
  - Rambam Health Care Campus, Haifa
  - Sheba Medical Center, Ramat Gan
  - Assuta Medical Centers, Tel Aviv
  - Tel Aviv Sourasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No